CLINICAL TRIAL: NCT05183425
Title: The Exploratory Study of Patient-derived Organoids for the Prediction and Evaluation of Clinical Efficiency Effect of Colorectal Cancer Liver Metastasis
Brief Title: Patient-derived Organoids Predicts the Clinical Efficiency of Colorectal Liver Metastasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhang, Director of the department of colorectal surgery, Changhai Hospital
Other Study IDs: CHCS-PDO
Record Dates: First submitted 2021-12-26; First posted 2022-01-10 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Explore the Consistency of Drug Sensitivity Between Primary Colorectal Cancer and Liver Metastases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Accumulating evidence indicates that patient- derived organoids (PDOs) can predict drug responses in the clinic. Metastasis is the main cause of death in colorectal cancer patients, and the treatment of patients with liver metastasis remains poor. Tumor heterogeneity is the cause of treatment failure. In this study, we aim the investigate the consistency of drug sensitivity for the matched primary and metastatic tumor in patients with liver metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven colorectal cancer with liver metastasis
* Aged between 18 and 70 years
* Written informed and signed consent
* Accessible to surgery sample of metastasis and primary tumor

Exclusion Criteria:

* Less than 18 years and older than 70 years
* Not able to give informed consent
* Not accessible to surgery sample

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with histologically proven colorectal cancer with liver metastasis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The consistency of drug sensitivity | 3 years
  To test the consistency of drug sensitivity of primary tumor and its matched liver metastasis

SECONDARY OUTCOMES:
The establishment of PDO | 3 years
  To test the rate of PDO derived from primary and matched metastatic colorectal cancer .

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Colorectal Surgery in Changhai Hospital, Shanghai, Shanghai Municipality, China